## STASTICAL ANALYSIS PLAN AND RESULTS

**Project Title**: Reducing Spread of COVID-19 in a University Community Setting: Role of a Low-Cost Reusable Form-Fitting Fabric Mask

NCT Number: NCT04979858

#### STATISTICAL ANALYSIS PLAN

The proposed statistical analysis will include the use of single-factor ANOVA test to assess the importance of the various factors associated with the design of the Focal Mask (the Treatment) that would impact its performance in reducing the spread of COVID-19, which is caused by the SARS-CoV-2 virus. The Bonferroni t-test will be conducted *post hoc* to assess the statistical significance of the various factors.

#### **RESULTS OF THE STATISTICAL ANALYSIS**

We present the details of the statistical analysis of the 200 post-study survey responses received at the end of the clinical trial. A copy of the survey is given in Appendix I.

As shown in the post-study instrument in Appendix I, the subjects were asked to identify all the devices used during the six-week study, viz., surgical mask, N95, KN95, fabric mask, and Focal Mask (the Low-Cost Reusable Form-Fitting Fabric Mask given only to those in the Treatment group). All the subjects were then asked to rank their experiences with each of these devices during the study based on specific characteristics reflecting the key user requirements for a mask defined in earlier research and shown in Table 1 (Park and Jayaraman, 2020<sup>1</sup>).

-

<sup>&</sup>lt;sup>1</sup> Park, S., and Jayaraman, S., (2020) From containment to harm reduction from SARS-CoV-2: a fabric mask for enhanced effectiveness, comfort, and compliance, <u>The Journal of The Textile</u> Institute, 112:7, 1144-1158, DOI: 10.1080/00405000.2020.1805971.

Table 1. Performance requirements for masks

| Functionality | <ul> <li>Provide a barrier against transfer of</li> <li>Microorganisms</li> <li>Body Fluids</li> </ul> |
|---|---|
| Usability | <ul> <li>Particulate Material</li> <li>Breathable</li> <li>Odor-free</li> <li>Ease of Donning and Doffing</li> <li>Minimal Impact on Job Performance</li> <li>Does not impair communication</li> </ul> |
| Wearability | <ul><li>Lightweight</li><li>Comfortable</li><li>Soft on Skin</li></ul> |
| Shape Conformability | <ul> <li>Conform to Desired Facial Shape</li> <li>Customizable</li> <li>Dimensional Stability even after Multiple Launderings</li> </ul> |
| Durability | <ul> <li>Reusable Multiple Times</li> <li>Strong</li> <li>Does not Tear</li> </ul> |
| Maintainability | Ease of Care including Ease of Decontamination Ease of Laundering |
| Manufacturability | Ease of Fabrication Compatible with Standard Sewing Machines |
| Affordability | Material Cost Homemade (so, manufacturing cost is not considered) |
| Aesthetics | Aesthetically Pleasing Multiple Colors and Designs |

These user requirements drove the design and development of the Focal Mask. As seen in Table 1, the most important user need is that the mask must serve as a barrier against the transfer of microorganisms, body fluids (e.g., saliva, mucus), and particulate materials from the wearer to the outside. The mask must be breathable so that the user is comfortable during extended use. The mask must be odor-free because it will be worn for long periods of time. Since the mask is intended for public use including children and the elderly, it must be easy to don and doff and not require any special training to learn to use. When used in a workplace setting, it should not impair the wearer's communication, which might impact job performance. If it muffles or muzzles the sound from going out during speaking, the wearer will remove the mask from the mouth thereby defeating the very reason for wearing a mask. The mask must be lightweight, soft, and conform to the wearer's facial profile. It must be easy to decontaminate at home by laundering so that it can be reused. It should have dimensional stability, i.e., retain its shape and

size, after multiple launderings so that it remains effective. Masks are becoming an essential accessory in everyone's wardrobe. Individuals express themselves through their clothing – the designs, colors, fit, style, and so on. Therefore, the masks should be aesthetically pleasing so that individuals are less self-conscious when wearing them.

The 200 post-study responses from the subjects were analyzed along the following lines:

- Features of the masks including Focal Mask
- Impact of masks on performance/interactions in school and/or at work
- Impact of masks on social life and interactions
- Opinions on masking practices
- Recommendations on improving the Focal mask

#### **Features of the Masks including Focal Mask**

For each question, e.g., "The mask was breathable," the response data was aggregated for each mask type based on the ranking assigned by the subject on a 1-5 scale (1 – best and 5 – worst). The next step was to carry out statistical analysis to test whether the rankings by the subjects shown were indeed statistically different. Therefore, a single factor ANOVA test was carried out on the data to see if there were any significant differences in the responses for all the masks used.

#### **Breathability**

We use "breathability" to explain the statistical analysis methodology in detail. Table 2 shows the summary of responses for the breathability question.

| Breathability | | Ma | ask Type | | |
|---------------|------------|---------------|----------|------|-------------|
| breathability | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
| Count | 100 | 155 | 23 | 43 | 134 |
| Average | 1.9 | 1.8 | 2.6 | 2.4 | 2.3 |
| Mode | 2 | 1 | 3 | 3 | 3 |
| Median | 2 | 2 | 3 | 2 | 2 |
| SD | 0.85 | 0.83 | 1.16 | 1.14 | 1.05 |

Table 2. Summary of Responses for Breathability of Mask

In the table, count represents the number of responses ranking that specific mask. For instance, since the Focal mask was given only to the 100 subjects in the Treatment group, the count is 100. The count of 155 in surgical mask represents the number of subjects who used the surgical mask

during the six-week study. Likewise, 23 subjects reported using N95, 43 using KN95, and 134 using fabric mask, respectively. The average represents the computed average of the individual ranks assigned by the subjects for each mask. On the 1-5 scale rating, the lower the number better the perceived performance. For instance, in Table 2, the surgical mask scored 1.8 in comparison to the Focal Mask with a score of 1.9, N95 with a score of 2.6, KN95 with 2.4, and fabric mask with 2.3, respectively. The mode and median rankings for each mask are also shown in the table. Figure 1 shows a graphical representation of the ranking of responses for the different masks in Table 2.



Figure 1. Ranking of Breathability of Masks Used by Subjects in the Study

**Statistical Analysis**: The next step was to test whether the rankings by the subjects shown in the figure (and table) were indeed statistically different. Therefore, a single factor ANOVA test was carried out on the data to see if there were any significant differences in the responses for all the masks used. Table 3 shows the result of the ANOVA test.

Table 3. Summary of Single Factor ANOVA Test for Breathability of Masks

| ANOVA: Single Factor | | | | | | | |
|---|---|---|---|---|---|---|---|
| SUMMARY | | | | | | | |
| Groups | Count | Sum | | Average | Variance | | |
| Focal Mask | 100 | | 187 | 1.87 | 0.72030303 | | |
| Surgical Mask | 155 | | 274 | 1.7677419 | 0.685965647 | | |
| N95 | 23 | | 60 | 2.6086957 | 1.339920949 | | |
| KN95 | 43 | | 104 | 2.4186047 | 1.296788483 | | |
| Fabric Mask | 134 | | 314 | 2.3432836 | 1.099315453 | | |
| ANOVA | | | | | Significant | | |
| Source of Variation | SS | df | | MS | F | P-value | F crit |
| Between Groups | 40.0506063 | | 4 | 10.012652 | 11.0677516 | 1.43228E-08 | 2.391758 |
| Within Groups | 407.101042 | | 450 | 0.904669 | | | |
| Total | 447.1516484 | | 454 | | | | |

A comparison of the F and  $F_{crit}$  values in Table 3 shows that the difference is significant since F is greater than  $F_{crit}$ . Therefore, a post-hoc Bonferroni t-test was performed using a correction factor of 0.005 assuming equal variances in the two types (e.g., Focal Mask and surgical mask) for all mask types using the following two hypotheses:

**Null hypothesis**: There is no significant difference in the assessment of that specific performance parameter, e.g., breathability in this example, between the two different masks. **Alternate hypothesis**: There is a significant difference in the assessment of that specific performance parameter, e.g., breathability in this example, between the two different masks.

Table 4 provides a summary of the post-hoc Bonferroni t-test for breathability.

Table 4. Summary of Bonferroni Post Hoc t-test for Breathability

| Bonferroni Post Hoc Test (t-test) | | Bonferro | ni correction: |
|---|---|---|---|
| t-Test: Two-Sample Assuming Equal | Variances | | |
| Comparison | p Value | Hypothesis | |
| Focal Mask vs Surgical Mask | 0.341347658 | Null | |
| Focal Mask vs N95 | 0.000652144 | Alternate | |
| Focal Mask vs KN95 | 0.001780898 | Alternate | |
| Focal Mask vs Fabric Mask | 0.000270484 | Alternate | |
| Surgical Mask vs N95 | 2.8793E-05 | Alternate | |
| Surgical Mask vs KN95 | 4.42331E-05 | Alternate | |
| Surgical Mask vs Fabric Mask | 3.63761E-07 | Alternate | |
| N95 vs KN95 | 0.522832795 | Null | |
| N95 vs Fabric Mask | 0.271069012 | Null | |
| KN95 vs Fabric Mask | 0.688674797 | Null | |

The table shows the applicable hypothesis (Null or Alternate) for each comparison based on the p value indicating whether the difference in breathability is statistically significant or not. Since the null hypothesis is applicable, there is no significant difference between the breathability of the Focal Mask and the surgical mask. However, the Focal Mask is significantly better than that of all the other mask types because the Alternate hypothesis is applicable. The breathability of the surgical mask is also significantly better than that of the other masks.

In a similar manner, the responses for the other questions (from Q2 through Q12 in the post-study survey) were analyzed. The results from the statistical analysis along the lines of Tables 2 through 4 are shown in Appendix II.

Table 5 shows the summary of the hypotheses applicable to each parameter assessed for all the masks used by the subjects in the post-study survey. It shows the assessment of the Focal Mask in comparison to the other masks used by the subjects during the study. It is important to note that the Focal Mask was given only to the 100 subjects in the Treatment group.

Table 5. Assessment of Focal Mask with respect to the other masks used by the subjects

| | Focal Mask | Focal Mask | Focal Mask | Focal Mask | Surgical Mask | Surgical Mask | Surgical Mask | N95 | N95 | KN95 |
|---|---|---|---|---|---|---|---|---|---|---|
| Comparison | vs | VS | VS | VS | vs | vs | vs | VS | VS | vs |
| · | Surgical Mask | N95 | KN95 | Fabric Mask | N95 | KN95 | Fabric Mask | KN95 | Fabric | Fabric |
| Q1. The mask was breathable | Null | Alternate | Alternate | Alternate | Alternate | Alternate | Alternate | Null | Null | Null |
| Q2. The mask conformed to the shape of my face to prevent leakage | Alternate | Alternate | Alternate | Alternate | Alternate | Alternate | Alternate | Null | Null | Alternate |
| Q3. The mask stayed in place when speaking to others | Alternate | Alternate | Alternate | Alternate | Null | Null | Null | Null | Null | Null |
| Q4. The mask did not require me to speak louder to others for them to hear me | Null | Alternate | Alternate | Alternate | Null | Alternate | Alternate | Null | Null | Null |
| Q5. The mask was easy to put on | Alternate | Alternate | Alternate | Alternate | Alternate | Alternate | Alternate | Null | Null | Null |
| Q6. The mask was easy to take off | Alternate | Alternate | Alternate | Alternate | Alternate | Alternate | Alternate | Null | Null | Null |
| Q7. The mask was comfortable to wear | Null | Null | Null | Null | Alternate | Null | Null | Null | Alternate | Null |
| Q8. The mask was soft on my skin | Alternate | Alternate | Alternate | Alternate | Null | Null | Alternate | Null | Alternate | Alternate |
| Q9. The mask did not cause rashes on my face | | | | | Null | | | | | |
| Q10. The mask did not leave traces or marks on my face during continuous use | Alternate | Null | Null | Alternate | Alternate | Alternate | Null | Null | Alternate | Alternate |
| Q11. The mask stayed away from my lips when I had it on | Alternate | Null | Null | Alternate | Null | Alternate | Null | Null | Null | Alternate |
| Q12. The mask did not have an odor to it when I wore it | Null | Null | Null | Alternate | Null | Null | Alternate | Null | Null | Null |

#### RESULTS AND ANALYSIS PERTAINING TO THE PRIMARY AIM

The primary aim of the study has been to test the role of the newly developed reusable form-fitting fabric mask, viz., the Focal Mask, in reducing the spread of COVID-19 in a community setting comprising undergraduate students living in dormitories at Georgia Tech.

Simulating a "Real" Community Setting: One of the key features of the study has been to simulate a "real" community setting in which individual behaviors cannot be specified, monitored, or controlled. Therefore, regular health diagnostic testing for COVID-19 was not mandated for the subjects in the study. In this effort to simulate a real community setting, it is acknowledged that subjects who became infected, but were asymptomatic, would not have been tested; as a result, there was a potential for undercounting the number of positive cases during the study. Likewise, during the study, instead of being required to wear a specific type of mask, the subjects were free to use the type of mask they preferred except for those selected to be in the Treatment group in which case they were required to use the Focal Mask (the Low-Cost Reusable Form-Fitting Fabric Mask) during the two-week Treatment phase.

#### **Health Diagnostic Testing**

Table 6 shows the health diagnostic testing for COVID-19 reported by subjects in the study during the three phases, viz., Pre-Treatment, Treatment, and Post-Treatment, respectively. This is based on the analysis of the 8,335 responses from the daily surveys from subjects enrolled in the Study. At the beginning of the study, there were 201 subjects. One subject withdrew from the study in accordance with the IRB-approved protocol for having tested positive on the seventh day of the Pre-Treatment phase of the study.

Table 6. Health Diagnostic Testing for COVID-19

| | Dro Tr | eatment | Troa | tment | Post Tr | eatment |
|---|---|---|---|---|---|---|
| Number of Subjects | Pie-iii | eaument | Hea | unent | PUSI-11 | eaument |
| | Control | Treatment | Control | Treatment | Control | Treatment |
| Who tested at least once | 69 | 77 | 72 | 82 | 61 | 67 |
| Who did not test | 32 | 23 | 28 | 18 | 39 | 33 |
| With Symptoms | 43 | 52 | 46 | 38 | 41 | 27 |
| , ' ' | | | _ | | | |
| Tested with Symptoms | 26 | 35 | 35 | 28 | 24 | 18 |
| Without Symptoms | 58 | 48 | 54 | 62 | 59 | 73 |
| Tested without Symptoms | 43 | 42 | 37 | 54 | 37 | 49 |
| | - | | | | | |
| Duamatian of Cubicata | Pre-Treatment | | Treatment | | Post-Treatment | |
| Propotion of Subjects | Control | Treatment | Control | Treatment | Control | Treatment |
| Who tested at least once | 68% | 77% | 72% | 82% | 61% | 67% |
| Who did not test | 32% | 23% | 28% | 18% | 39% | 33% |
| | 1 | | ı | T | ı | |
| With symptoms who tested | 60% | 67% | 76% | 74% | 59% | 67% |
| Without symptoms who tested | 74% | 88% | 69% | 87% | 63% | 67% |

As seen in the table and in Figure 2, a majority of the students in both groups (Control and Treatment) tested at least once in each phase of the three-phase study. Moreover, a majority of the students with symptoms tested in both groups in all three phases. Routine testing, i.e., testing that is voluntary and not triggered by symptoms is also high, ranging from 63% in the Post-treatment Control group to 88% in the Pre-treatment Treatment group.



Figure 2. Symptom-driven testing and routine testing in subject population.

One of the key objectives of the study was to simulate a "real" community setting in which individual behaviors cannot be specified, monitored, or controlled. So, regular testing was not

mandated for the subjects in the study. Figures 2 and 3 show the behavior of subjects in the chosen university community setting. Overall, 91% of the subjects underwent testing during the six weeks while 9% chose not to test during the entire six weeks of the study.



Figure 3. COVID-19 Testing in Subject Population during Six Weeks of Study

#### **COVID-19 Infections during Study Period: Georgia Tech and Subject Population**

Table 7 shows the results of COVID-19 saliva tests conducted on campus in the Georgia Tech population during the six weeks of the study. The days corresponding to the three phases of the study (Pre-Treatment, Treatment, and Post-Treatment) are highlighted in different colors.

Table 7. Georgia Tech COVID-19 Test Data

| Dayin | | Number | Number of | Po | sitivity by Loc | cation |
|---|---|---|---|---|---|---|
| Day in<br>Study | Date | of Positive | Tests | Greek | Residence | Off-Campus |
| Study | | Individuals | Conducted | House | Hall | Student |
| 1 | 9/10/2021 | 29 | 3019 | 2 | 12 | 13 |
| 2 | 9/11/2021 | 15 | 1412 | 2 | 7 | 5 |
| 3 | 9/12/2021 | 2 | 0 | 0 | 1 | 0 |
| 4 | 9/13/2021 | 2 | 585 | 0 | 0 | 0 |
| 5 | 9/14/2021 | 7 | 1423 | 1 | 1 | 3 |
| 6 | 9/15/2021 | 5 | 1842 | 0 | 1 | 1 |
| 7 | 9/16/2021 | 13 | 1484 | 1 | 6 | 4 |
| 8 | 9/17/2021 | 5 | 1666 | 0 | 2 | 1 |
| 9 | 9/18/2021 | 10 | 932 | 1 | 4 | 4 |
| 10 | 9/19/2021 | 1 | 1 | 0 | 0 | 1 |
| 11 | 9/20/2021 | 4 | 598 | 0 | 1 | 1 |
| 12 | 9/21/2021 | 7 | 979 | 0 | 2 | 4 |

| 13 9/22/2021 5 1954 1 2 2 14 9/23/2021 8 1395 0 1 4 15 9/24/2021 1 43 0 0 1 16 9/25/2021 12 2365 1 4 4 17 9/26/2021 2 1 0 1 0 18 9/27/2021 6 592 0 2 3 19 9/28/2021 7 973 1 1 3 20 9/29/2021 2 2126 1 0 1 21 9/30/2021 5 1389 0 1 4 22 10/1/2021 4 778 0 0 3 23 10/2/2021 5 960 0 2 2 24 10/3/2021 2 0 0 0 0 |
|---|
| 15 9/24/2021 1 43 0 0 1 16 9/25/2021 12 2365 1 4 4 17 9/26/2021 2 1 0 1 0 18 9/27/2021 6 592 0 2 3 19 9/28/2021 7 973 1 1 3 20 9/29/2021 2 2126 1 0 1 21 9/30/2021 5 1389 0 1 4 22 10/1/2021 4 778 0 0 3 23 10/2/2021 5 960 0 2 2 24 10/3/2021 2 0 0 0 0 |
| 16 9/25/2021 12 2365 1 4 4 17 9/26/2021 2 1 0 1 0 18 9/27/2021 6 592 0 2 3 19 9/28/2021 7 973 1 1 3 20 9/29/2021 2 2126 1 0 1 21 9/30/2021 5 1389 0 1 4 22 10/1/2021 4 778 0 0 3 23 10/2/2021 5 960 0 2 2 24 10/3/2021 2 0 0 0 0 |
| 17 9/26/2021 2 1 0 1 0 18 9/27/2021 6 592 0 2 3 19 9/28/2021 7 973 1 1 3 20 9/29/2021 2 2126 1 0 1 21 9/30/2021 5 1389 0 1 4 22 10/1/2021 4 778 0 0 3 23 10/2/2021 5 960 0 2 2 24 10/3/2021 2 0 0 0 0 |
| 18 9/27/2021 6 592 0 2 3 19 9/28/2021 7 973 1 1 3 20 9/29/2021 2 2126 1 0 1 21 9/30/2021 5 1389 0 1 4 22 10/1/2021 4 778 0 0 3 23 10/2/2021 5 960 0 2 2 24 10/3/2021 2 0 0 0 0 |
| 19 9/28/2021 7 973 1 1 3 20 9/29/2021 2 2126 1 0 1 21 9/30/2021 5 1389 0 1 4 22 10/1/2021 4 778 0 0 3 23 10/2/2021 5 960 0 2 2 24 10/3/2021 2 0 0 0 0 |
| 20 9/29/2021 2 2126 1 0 1 21 9/30/2021 5 1389 0 1 4 22 10/1/2021 4 778 0 0 3 23 10/2/2021 5 960 0 2 2 24 10/3/2021 2 0 0 0 0 |
| 21 9/30/2021 5 1389 0 1 4 22 10/1/2021 4 778 0 0 3 23 10/2/2021 5 960 0 2 2 24 10/3/2021 2 0 0 0 0 |
| 22 10/1/2021 4 778 0 0 3 23 10/2/2021 5 960 0 2 2 24 10/3/2021 2 0 0 0 0 |
| 23 10/2/2021 5 960 0 2 2 24 10/3/2021 2 0 0 0 0 |
| 24 10/3/2021 2 0 0 0 0 |
| 25 40/4/2024 2 544 2 2 |
| 25 10/4/2021 3 541 0 2 0 |
| 26 10/5/2021 4 1014 0 2 1 |
| 27 10/6/2021 6 1554 0 1 2 |
| 28 10/7/2021 1 1376 0 1 0 |
| 29 10/8/2021 2 281 0 0 0 |
| 30 10/9/2021 0 1932 0 0 0 |
| 31 10/10/2021 6 51 0 2 2 |
| 32 10/11/2021 2 51 0 0 1 |
| 33 10/12/2021 0 495 0 0 0 |
| 34 10/13/2021 3 577 1 0 1 |
| 35 10/14/2021 2 1852 0 0 2 |
| 36 10/15/2021 6 1891 1 0 4 |
| 37 10/16/2021 1 47 0 0 1 |
| 38 10/17/2021 0 0 0 0 0 |
| 39 10/18/2021 0 557 0 0 0 |
| 40 10/19/2021 1 960 0 0 1 |
| 41 10/20/2021 5 1470 0 1 4 |
| 42 10/21/2021 0 1171 0 0 0 |

As seen in the table, while the number of positive cases in the general campus population is low, individuals are testing positive for COVID-19. It is important to note that no data was collected on the masking practices of the Georgia Tech population that got tested during the period. In contrast, none of the subjects reported testing positive in the daily surveys during the six weeks of the study. Typically when subjects experienced symptoms, they got tested (Figure 2). However, subjects who were infected, but were asymptomatic, did not get tested because testing was not mandatory for participation in the study since one of the goals was to simulate a "real" community setting. It is acknowledged that there was a potential for undercounting the number of positive cases in the subject population during the study.

#### **CONCLUSIONS**

We draw on the preceding findings and analysis to present the following major conclusions from the study:

- An IRB-approved clinical trial to test the effectiveness of a prototype low-cost reusable form-fitting fabric mask (Focal Mask) to reduce infectious disease spread, i.e., COVID-19, through respiratory secretions in undergraduate students living in dormitories at Georgia Tech was completely successfully. This subject population (201) was chosen due to the significant person-to-person contact that occurs in residences, classes, and social activities among university students.
- To simulate a "real" community setting in which individual behaviors cannot be specified, monitored, or controlled, regular health diagnostic testing for COVID-19 during the study was not mandated for the subjects.
  - In this effort to simulate a real community setting, it is acknowledged that subjects who became infected, but were asymptomatic, would not have been tested; as a result, there is a potential for undercounting the number of reported positive cases during the study.
  - Likewise, during the study, instead of being required to wear a specific type of mask, the subjects were free to use the type of mask they preferred except for those selected to be in the Treatment group in which case they were required to use the Focal Mask during the two-week Treatment phase.
- Apart from the one positive COVID-19 transmission reported by a subject on Day Seven of the study (Pre-Treatment phase), no confirmed positive COVID-19 transmission was reported during the six weeks of the study. The subject who reported testing positive had been quarantining from Day One of the study due to exposure to an infected individual; the subject withdrew in accordance with the IRB-approved study protocol.
- In contrast, during the same six-week period of the study, Georgia Tech's COVID-19 testing data showed positive COVID-19 cases in the student population. It is important to note that no data was collected on the masking practices of the Georgia Tech population that got tested during the period.
- All the subjects reported that they wore their masks when in public during the day, which is one of the key preventative measures to reduce the spread of COVID-19.
- Despite the high degrees of interaction reported by the subjects (in residence halls, in classes, during group meetings, during dining, and in social settings), the use of masks, including the Focal Mask, could have served as one of the preventative measures to prevent the spread of COVID-19 in the subject population. It is important to reiterate that regular testing for COVID-19 was not mandated for the subjects

- during the study; consequently, subjects who were infected, but were asymptomatic, would not have been counted.
- The design and structure of the Focal Mask, including having a built-in filter, have been validated from the viewpoint of the various user requirements including breathability, shape conformability, speech intelligibility, and comfort, among others.

In closing, wearing a mask, such as the prototype Focal Mask, could be an effective tool as one of the preventative measures to prevent the spread of infectious diseases, such as COVID-19, through respiratory secretion in a community setting with a high degree of interaction among individuals living in university residence halls. The overwhelming willingness of the subject population to wear masks as a means to control the spread of infection was an important factor in the transmission rates observed in the study population.

Appendix I: Post-Study Survey

# **Post-Study Questionnaire Treatment**

| Start of Bloc | k: Intro |
|---|---|
| 1 Thank you f | or your diligent participation in this important Study! This is the last Survey!! |
| want to learn | arn about your experience with masks you have used during the Study. We also about your views on using masks in public and in social settings. We want you to ur total experience during the Study and complete this Survey. |
| Please compl | ete this Survey by <b>4:59 p.m. on Tuesday, October 26th.</b> |
| End of Block | : Intro |
| Start of Bloc | k: Post-Study Survey |
| Select all mas | sks you used during the Study: |
| | Focal Fabric Mask (5) |
| | Surgical Mask (1) |
| | N-95 Respirator (2) |
| | KN-95 Respirator (3) |
| | Fabric Mask (4) |
| Page Break | |

Rate the performance of each mask you used in the following categories.

Scale: 1 - best; 5 - worst.

If the performance is similar, you can provide the same rating. Check "Not Applicable" if you did not use that mask.

The mask was breathable.

Best Worst

1 2 3 4 5

Focal Mask ()

Surgical Mask ()

N95 ()

KN95 ()

Fabric Mask ()

The mask conformed to the shape of my face to prevent leakage.

Best

Not Applicable Worst

1 2 3 4 5

Focal Mask ()

Surgical Mask ()

N95 ()

KN95 ()

Fabric Mask ()

| The mask stayed in place when speaking to othe | ers.<br>Best | | | Not App | licable 🗌<br>Worst |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 |
| Focal Mask () | | | - | | - |
| Surgical Mask () | | | - | | = |
| N95 () | | | - | | = |
| KN95 () | | | | | = |
| Fabric Mask () | | | - | | = |

The mask was easy to put on.

Best Worst

1 2 3 4 5

Focal Mask ()

Surgical Mask ()

N95 ()

KN95 ()

Fabric Mask ()

The mask was easy to take off.

Best Worst

1 2 3 4 5

Focal Mask ()

Surgical Mask ()

N95 ()

KN95 ()

Fabric Mask ()

The mask was comfortable to wear.

Best Worst

1 2 3 4 5

Focal Mask ()

Surgical Mask ()

N95 ()

KN95 ()

Fabric Mask ()

| The mask was soft on my skin. | Best | | | Not App | licable<br>Worst |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 |
| Focal Mask () | | | - | | - |
| Surgical Mask () | | | - | | |
| N95 () | | | - | | - |
| KN95 () | | | - | | - |
| Fabric Mask () | | | <b>-</b> - | | - |

The mask did not cause rashes on my face.

Best Worst

1 2 3 4 5

Focal Mask ()

Surgical Mask ()

N95 ()

KN95 ()

Fabric Mask ()



The mask stayed away from my lips when I had it on.

Best

Not Applicable 
Worst

1 2 3 4 5

Focal Mask ()

Surgical Mask ()

N95 ()

KN95 ()

Fabric Mask ()

The mask did not have an odor to it when I wore it.

Best

Tocal Mask ()

Surgical Mask ()

Not Applicable Worst

1 2 3 4 5

Focal Mask ()

Ny5 ()

KN95 ()

Fabric Mask ()

Rate the washing performance of each mask you used.

Scale: 1 - best; 5 - worst.

If the performance is similar, you can provide the same rating. Check "Not Applicable" if you did not use that type of mask or is not washable (e.g., Surgical mask).

| The mask was easy to wash. | Best<br>1 | 2 | 2 | Not App | licable 🗌<br>Worst<br>5 |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 |
| Focal Mask () | | | - | | - |
| Surgical Mask () | | | | | - |
| N95 () | | | - | | |
| KN95 () | | | - | | - |
| Fabric Mask () | | | - | | - |
| The mask did not change its shape or fit after it v | was wash<br>Best | ned. | | Not App | licable Worst |
| The mask did not change its shape or fit after it v | | ned.<br>2 | 3 | Not App | |
| The mask did not change its shape or fit after it version of the shape | Best | | 3 | | Worst |
| | Best | | 3 | | Worst |
| Focal Mask () | Best | | 3 | | Worst |
| Focal Mask () Surgical Mask () | Best | | 3 | | Worst |
| Focal Mask () Surgical Mask () N95 () | Best | | 3 | | Worst |

The mask did not develop a bad odor after it was used and washed a few times. Not Applicable **Best** Worst 1 2 3 5 4 Focal Mask () Surgical Mask () N95 () KN95 () Fabric Mask () Wearing the mask impeded my performance in class or at my work. O Strongly agree (1) O Somewhat agree (2) O Neither agree nor disagree (3) O Somewhat disagree (4) Strongly disagree (5) Wearing the mask limited my social life. O Strongly agree (1) O Somewhat agree (2) O Neither agree nor disagree (3) O Somewhat disagree (4) Strongly disagree (5)

| O Strongly agree (1) | | | | | |
|---|---|---|---|---|---|
| O Somewl | hat agree (2) | | | | |
| O Neither agree nor disagree (3) | | | | | |
| ○ Somewhat disagree(4) | | | | | |
| | disagree (5) | | | | |
| _ | e <i>color</i> of my ma | | | I / Formal clothin | g is very |
| important to me | e. Fill out accordir | | v.<br>Neither agree | | |
| | Strongly<br>agree (12) | Somewhat<br>agree (13) | nor disagree<br>(14) | Somewhat<br>disagree (15) | Strongly<br>disagree (16) |
| School<br>(Casual) (11) | 0 | 0 | 0 | 0 | 0 |
| Social (Semi-<br>formal) (12) | 0 | 0 | 0 | 0 | $\circ$ |
| Business<br>(Formal) (13) | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| - | e <b>des<i>ign (patter</i><br/>nt</b> to me. Fill out a | | each row. | / Semi-formal / F | <u>formal</u> clothing |
| | Strongly<br>agree (12) | Somewhat agree (13) | Neither agree<br>nor disagree<br>(14) | Somewhat disagree (15) | Strongly<br>disagree (16) |
| School<br>(Casual) (11) | 0 | 0 | 0 | 0 | 0 |
| Social (Semi-<br>formal) (12) | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Business<br>(Formal) (13) | 0 | $\circ$ | 0 | 0 | $\circ$ |

I had reservations about wearing the mask when meeting socially with my friends.

Coordinating the *style* of my mask with my <u>Casual / Semi-formal / Formal</u> clothing is very important to me. Fill out accordingly for each row.

| | Strongly<br>agree (12) | Somewhat agree (13) | Neither agree<br>nor disagree<br>(14) | Somewhat<br>disagree (15) | Strongly<br>disagree (16) |
|---|---|---|---|---|---|
| School<br>(Casual) (11) | 0 | 0 | 0 | 0 | 0 |
| Social (Semi-<br>formal) (12) | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Business<br>(Formal) (13) | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| <ul><li>Strongly</li><li>Somew</li><li>Neither</li><li>Somew</li></ul> | one should wear more agree (1) hat agree (2) agree nor disagre hat disagree (4) or disagree (5) | | public settings. | | |
| Strongly Somew Neither Somew | one should wear more agree (1) hat agree (2) agree nor disagre hat disagree (4) or disagree (5) | | or public settings. | | |

| The reusability of the mask is important to me. |
|---|
| O Strongly agree (1) |
| O Somewhat agree (2) |
| O Neither agree nor disagree (3) |
| ○ Somewhat disagree (4) |
| O Strongly disagree (5) |
| Having a built-in filter is important to me. |
| ○ Strongly agree (1) |
| ○ Somewhat agree (2) |
| O Neither agree nor disagree (3) |
| ○ Somewhat disagree (4) |
| ○ Strongly disagree (5) |
| List any specific issues when wearing the focal mask. |
| What changes would you make to the design of the focal mask? |
| List any additional thoughts or input you have on your experience using the focal mask. |

# Appendix II: Statistical Analysis of Post-Study Surveys

# Q1. The mask was breathable.

**DATA: Summary** 

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 100 | 155 | 23 | 43 | 134 |
| Average | 1.9 | 1.8 | 2.6 | 2.4 | 2.3 |
| Mode | 2 | 1 | 3 | 3 | 3 |
| Median | 2 | 2 | 3 | 2 | 2 |
| SD | 0.85 | 0.83 | 1.16 | 1.14 | 1.05 |

## **ANOVA: Single Factor**

**SUMMARY** 

| Groups | Count | Sum | Average | Variance |
|---------------|-------|-----|-----------|-------------|
| Focal Mask | 100 | 187 | 1.87 | 0.72030303 |
| Surgical Mask | 155 | 274 | 1.7677419 | 0.685965647 |
| N95 | 23 | 60 | 2.6086957 | 1.339920949 |
| KN95 | 43 | 104 | 2.4186047 | 1.296788483 |
| Fabric Mask | 134 | 314 | 2.3432836 | 1.099315453 |

| ANOVA | | | | Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 40.0506063 | 4 | 10.012652 | 11.0677516 | 1.43228E-08 | 2.391758 |
| Within Groups | 407.101042 | 450 | 0.904669 | | | |
| Total | 447.1516484 | 454 | | | | |

Bonferroni correction:

0.005

## **Bonferroni Post Hoc Test (t-test)**

| | P Value | Hypothesis |
|------------------------------|-------------|------------|
| Focal Mask vs Surgical Mask | 0.341347658 | Null |
| Focal Mask vs N95 | 0.000652144 | Alternate |
| Focal Mask vs KN95 | 0.001780898 | Alternate |
| Focal Mask vs Fabric Mask | 0.000270484 | Alternate |
| Surgical Mask vs N95 | 2.8793E-05 | Alternate |
| Surgical Mask vs KN95 | 4.42331E-05 | Alternate |
| Surgical Mask vs Fabric Mask | 3.63761E-07 | Alternate |
| N95 vs KN95 | 0.522832795 | Null |
| N95 vs Fabric Mask | 0.271069012 | Null |
| KN95 vs Fabric Mask | 0.688674797 | Null |

# Q2. The mask conformed to the shape of my face to prevent leakage.

#### **DATA: Summary**

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 100 | 156 | 25 | 42 | 133 |
| Average | 1.4 | 2.9 | 2.1 | 2.0 | 2.6 |
| Mode | 1 | 3 | 2 | 1 | 3 |
| Median | 1 | 3 | 2 | 2 | 3 |
| SD | 0.89 | 1.02 | 1.20 | 1.19 | 0.92 |

## **ANOVA: Single Factor**

**SUMMARY** 

| Groups | Count | Sum | Average | Variance |
|---------------|-------|-----|-----------|-------------|
| Focal Mask | 100 | 140 | 1.4 | 0.787878788 |
| Surgical Mask | 156 | 455 | 2.9166667 | 1.044623656 |
| N95 | 25 | 53 | 2.12 | 1.443333333 |
| KN95 | 42 | 84 | 2 | 1.414634146 |
| Fabric Mask | 133 | 343 | 2.5789474 | 0.851674641 |

| ANOVA | | | | Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 153.7569298 | 4 | 38.439232 | 38.9594649 | 5.05948E-28 | 2.391714 |
| Within Groups | 444.9777193 | 451 | 0.9866468 | | | |
| Total | 598.7346491 | 455 | | | | |

Bonferroni correction: 0.005

## **Bonferroni Post Hoc Test (t-test)**

| 2 1 2 2 2 1 1 2 2 2 2 2 2 2 2 2 2 2 2 2 | P Value | Hypothesis |
|-----------------------------------------|-------------|------------|
| Focal Mask vs Surgical Mask | 3.42742E-27 | Alternate |
| Focal Mask vs N95 | 0.00102224 | Alternate |
| Focal Mask vs KN95 | 0.001183617 | Alternate |
| Focal Mask vs Fabric Mask | 3.23802E-19 | Alternate |
| Surgical Mask vs N95 | 0.000530197 | Alternate |
| Surgical Mask vs KN95 | 1.40284E-06 | Alternate |
| Surgical Mask vs Fabric Mask | 0.003698606 | Alternate |
| N95 vs KN95 | 0.691992985 | Null |
| N95 vs Fabric Mask | 0.03164194 | Null |
| KN95 vs Fabric Mask | 0.001191605 | Alternate |

# Q3. The mask stayed in place when speaking to others.

#### **DATA: Summary**

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 100 | 158 | 23 | 39 | 136 |
| Average | 1.4 | 2.3 | 2.1 | 2.2 | 2.4 |
| Mode | 1 | 2 | 1 | 1 | 2 |
| Median | 1 | 2 | 2 | 2 | 2 |
| SD | 0.69 | 1.01 | 1.31 | 1.33 | 1.13 |

## **ANOVA: Single Factor**

**SUMMARY** 

| Groups | Count | Sum | Average | Variance |
|---------------|-------|-----|-----------|-------------|
| Focal Mask | 100 | 139 | 1.39 | 0.482727273 |
| Surgical Mask | 158 | 370 | 2.3417722 | 1.02894461 |
| N95 | 23 | 48 | 2.0869565 | 1.719367589 |
| KN95 | 39 | 84 | 2.1538462 | 1.765182186 |
| Fabric Mask | 136 | 331 | 2.4338235 | 1.284477124 |

| ANOVA | | | | Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 74.46353756 | 4 | 18.615884 | 17.21707438 | 3.73625E-13 | 2.391714 |
| Within Groups | 487.6417256 | 451 | 1.0812455 | | | |
| Total | 562.1052632 | 455 | | | | |

Bonferroni correction:

0.005

## **Bonferroni Post Hoc Test (t-test)**

| | P Value | Hypothesis |
|------------------------------|-------------|------------|
| Focal Mask vs Surgical Mask | 9.17549E-15 | Alternate |
| Focal Mask vs N95 | 0.000490665 | Alternate |
| Focal Mask vs KN95 | 2.00213E-05 | Alternate |
| Focal Mask vs Fabric Mask | 2.19623E-14 | Alternate |
| Surgical Mask vs N95 | 0.280765228 | Null |
| Surgical Mask vs KN95 | 0.332912844 | Null |
| Surgical Mask vs Fabric Mask | 0.463063617 | Null |
| N95 vs KN95 | 0.848066267 | Null |
| N95 vs Fabric Mask | 0.186638708 | Null |
| KN95 vs Fabric Mask | 0.192832634 | Null |

# Q4. The mask did not require me to speak louder to others for them to hear me

#### **DATA: Summary**

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 100 | 156 | 23 | 41 | 134 |
| Average | 1.9 | 2.0 | 2.6 | 2.6 | 2.6 |
| Mode | 2 | 2 | 2 | 2 | 3 |
| Median | 2 | 2 | 2 | 2 | 3 |
| SD | 0.84 | 1.00 | 1.23 | 1.20 | 1.14 |

## **ANOVA: Single Factor**

**SUMMARY** 

| Groups | Count | Sum | Average | Variance |
|---------------|-------|-----|-----------|-------------|
| Focal Mask | 100 | 189 | 1.89 | 0.704949495 |
| Surgical Mask | 156 | 308 | 1.974359 | 1.005789909 |
| N95 | 23 | 60 | 2.6086957 | 1.52173913 |
| KN95 | 41 | 106 | 2.5853659 | 1.448780488 |
| Fabric Mask | 134 | 349 | 2.6044776 | 1.293513635 |

| ANOVA | | | | Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 49.02198174 | 4 | 12.255495 | 11.24945286 | 1.04581E-08 | 2.391802 |
| Within Groups | 489.1542297 | 449 | 1.0894304 | | | |
| Total | 538.1762115 | 453 | | | | |

Bonferroni correction:

0.005

## **Bonferroni Post Hoc Test (t-test)**

| | P Value | Hypothesis |
|------------------------------|-------------|------------|
| Focal Mask vs Surgical Mask | 0.485432948 | Null |
| Focal Mask vs N95 | 0.001029174 | Alternate |
| Focal Mask vs KN95 | 0.000142949 | Alternate |
| Focal Mask vs Fabric Mask | 2.74912E-07 | Alternate |
| Surgical Mask vs N95 | 0.006662839 | Null |
| Surgical Mask vs KN95 | 0.001057963 | Alternate |
| Surgical Mask vs Fabric Mask | 9.35402E-07 | Alternate |
| N95 vs KN95 | 0.941451107 | Null |
| N95 vs Fabric Mask | 0.98707171 | Null |
| KN95 vs Fabric Mask | 0.926110828 | Null |

## Q5. The mask was easy to put on.

**DATA: Summary** 

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 100 | 156 | 20 | 40 | 134 |
| Average | 3.0 | 1.3 | 2.1 | 1.8 | 1.7 |
| Mode | 2 | 1 | 1 | 1 | 1 |
| Median | 3 | 1 | 1.5 | 1 | 1 |
| SD | 1.12 | 0.56 | 1.28 | 1.22 | 0.96 |

## **ANOVA: Single Factor**

**SUMMARY** 

| Groups | Count | Sum | Average | Variance |
|---------------|-------|-----|-----------|-------------|
| Focal Mask | 100 | 300 | 3 | 1.252525253 |
| Surgical Mask | 156 | 195 | 1.25 | 0.317741935 |
| N95 | 20 | 41 | 2.05 | 1.628947368 |
| KN95 | 40 | 73 | 1.825 | 1.481410256 |
| Fabric Mask | 134 | 223 | 1.6641791 | 0.916451577 |

| ANOVA | | | | Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 193.8613847 | 4 | 48.465346 | 56.18430455 | 2.37271E-38 | 2.391982 |
| Within Groups | 383.8630597 | 445 | 0.8626136 | | | |
| Total | 577.7244444 | 449 | | | | |

Bonferroni correction: 0.005

## **Bonferroni Post Hoc Test (t-test)**

| | P Value | Hypothesis |
|------------------------------|-------------|------------|
| Focal Mask vs Surgical Mask | 3.31868E-42 | Alternate |
| Focal Mask vs N95 | 0.000968692 | Alternate |
| Focal Mask vs KN95 | 2.02822E-07 | Alternate |
| Focal Mask vs Fabric Mask | 2.9672E-19 | Alternate |
| Surgical Mask vs N95 | 1.65668E-06 | Alternate |
| Surgical Mask vs KN95 | 2.03884E-05 | Alternate |
| Surgical Mask vs Fabric Mask | 7.51657E-06 | Alternate |
| N95 vs KN95 | 0.509151547 | Null |
| N95 vs Fabric Mask | 0.110550134 | Null |
| KN95 vs Fabric Mask | 0.383693557 | Null |

## Q6. The mask was easy to take off.

#### **DATA: Summary**

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 100 | 156 | 23 | 39 | 133 |
| Average | 2.9 | 1.2 | 2.0 | 1.6 | 1.5 |
| Mode | 3 | 1 | 1 | 1 | 1 |
| Median | 3 | 1 | 1 | 1 | 1 |
| SD | 1.15 | 0.46 | 1.40 | 1.11 | 0.86 |

## **ANOVA: Single Factor**

**SUMMARY** 

| Groups | Count | Sum | Average | | Variance |
|---------------|-------|-----|---------|-----------|-------------|
| Focal Mask | 100 | 2 | 294 | 2.94 | 1.32969697 |
| Surgical Mask | 156 | 1 | 186 | 1.1923077 | 0.207940447 |
| N95 | 23 | | 45 | 1.9565217 | 1.95256917 |
| KN95 | 39 | | 63 | 1.6153846 | 1.24291498 |
| Fabric Mask | 133 | 1 | 194 | 1.4586466 | 0.735019367 |

| ANOVA | | | | Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 202.9903368 | 4 | 50.747584 | 64.46787857 | 5.34744E-43 | 2.391936 |
| Within Groups | 351.0806166 | 446 | 0.7871763 | | | |
| Total | 554.0709534 | 450 | | | | |

Bonferroni correction: 0.005

## **Bonferroni Post Hoc Test (t-test)**

| | P Value | Hypothesis |
|------------------------------|-------------|------------|
| Focal Mask vs Surgical Mask | 9.54529E-44 | Alternate |
| Focal Mask vs N95 | 0.000568015 | Alternate |
| Focal Mask vs KN95 | 8.36193E-09 | Alternate |
| Focal Mask vs Fabric Mask | 1.07145E-23 | Alternate |
| Surgical Mask vs N95 | 4.32986E-07 | Alternate |
| Surgical Mask vs KN95 | 0.000299259 | Alternate |
| Surgical Mask vs Fabric Mask | 0.000876543 | Alternate |
| N95 vs KN95 | 0.294134953 | Null |
| N95 vs Fabric Mask | 0.022075933 | Null |
| KN95 vs Fabric Mask | 0.351426344 | Null |

# Q7. The mask was comfortable to wear.

**DATA: Summary** 

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 100 | 156 | 21 | 38 | 133 |
| Average | 2.2 | 2.1 | 2.8 | 2.5 | 2.1 |
| Mode | 1 | 2 | 3 | 3 | 2 |
| Median | 2 | 2 | 3 | 2.5 | 2 |
| SD | 1.12 | 0.94 | 1.36 | 0.83 | 1.00 |

## **ANOVA: Single Factor**

SUMMARY

| Groups | Count | Sum | Average | Variance |
|---------------|-------|-----|-----------|-------------|
| Focal Mask | 100 | 216 | 2.16 | 1.246868687 |
| Surgical Mask | 156 | 323 | 2.0705128 | 0.878866832 |
| N95 | 21 | 59 | 2.8095238 | 1.861904762 |
| KN95 | 38 | 94 | 2.4736842 | 0.688477952 |
| Fabric Mask | 133 | 274 | 2.0601504 | 0.996354523 |

| ANOVA | | | | Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 15.16756458 | 4 | 3.7918911 | 3.700873587 | 0.00562111 | 2.392073 |
| Within Groups | 453.8949354 | 443 | 1.0245935 | | | |
| Total | 469.0625 | 447 | | | | |

Bonferroni correction:

0.005

## **Bonferroni Post Hoc Test (t-test)**

| | P Value | Hypothesis |
|------------------------------|-------------|------------|
| Focal Mask vs Surgical Mask | 0.490260663 | Null |
| Focal Mask vs N95 | 0.021564178 | Null |
| Focal Mask vs KN95 | 0.118026976 | Null |
| Focal Mask vs Fabric Mask | 0.47344125 | Null |
| Surgical Mask vs N95 | 0.001667626 | Alternate |
| Surgical Mask vs KN95 | 0.01608225 | Null |
| Surgical Mask vs Fabric Mask | 0.927632253 | Null |
| N95 vs KN95 | 0.243879271 | Null |
| N95 vs Fabric Mask | 0.002886109 | Alternate |
| KN95 vs Fabric Mask | 0.020849209 | Null |

# Q8. The mask was soft on my skin.

**DATA: Summary** 

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 100 | 156 | 21 | 40 | 133 |
| Average | 1.5 | 2.4 | 3.1 | 2.6 | 1.8 |
| Mode | 1 | 2 | 2 | 2 | 1 |
| Median | 1 | 2 | 3 | 2.5 | 2 |
| SD | 0.72 | 1.00 | 1.37 | 0.98 | 0.97 |

## **ANOVA: Single Factor**

**SUMMARY** 

| Groups | Count | Sum Average | | Variance |
|---------------|-------|-------------|-----------|-------------|
| Focal Mask | 100 | 146 | 1.46 | 0.513535354 |
| Surgical Mask | 156 | 379 | 2.4294872 | 1.00789909 |
| N95 | 21 | 65 | 3.0952381 | 1.89047619 |
| KN95 | 40 | 104 | 2.6 | 0.964102564 |
| Fabric Mask | 133 | 243 | 1.8270677 | 0.947140579 |

| ANOVA | | | | Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 98.4613386 | 4 | 24.615335 | 26.88078439 | 5.41403E-20 | 2.391982 |
| Within Groups | 407.4964392 | 445 | 0.9157223 | | | |
| Total | 505.9577778 | 449 | | | | |

Bonferroni correction: 0.005

## **Bonferroni Post Hoc Test (t-test)**

| | P Value | Hypothesis |
|------------------------------|-------------|------------|
| Focal Mask vs Surgical Mask | 3.59738E-15 | Alternate |
| Focal Mask vs N95 | 1.61966E-12 | Alternate |
| Focal Mask vs KN95 | 3.83691E-12 | Alternate |
| Focal Mask vs Fabric Mask | 0.001683178 | Alternate |
| Surgical Mask vs N95 | 0.007185694 | Null |
| Surgical Mask vs KN95 | 0.336977521 | Null |
| Surgical Mask vs Fabric Mask | 4.70092E-07 | Alternate |
| N95 vs KN95 | 0.109374734 | Null |
| N95 vs Fabric Mask | 5.83862E-07 | Alternate |
| KN95 vs Fabric Mask | 1.93755E-05 | Alternate |

# Q9. The mask did not cause rashes on my face.

#### **DATA: Summary**

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 98 | 156 | 22 | 39 | 131 |
| Average | 1.5 | 1.5 | 2.0 | 1.6 | 1.5 |
| Mode | 1 | 1 | 1 | 1 | 1 |
| Median | 1 | 1 | 1 | 1 | 1 |
| SD | 0.98 | 0.86 | 1.36 | 0.99 | 1.05 |

## **ANOVA: Single Factor**

SUMMARY

| Groups | Count | Sum | | Average | Variance |
|---------------|-------|-----|-----|-----------|-------------|
| Focal Mask | 98 | | 146 | 1.4897959 | 0.953503051 |
| Surgical Mask | 156 | | 238 | 1.525641 | 0.74127378 |
| N95 | 22 | | 43 | 1.9545455 | 1.854978355 |
| KN95 | 39 | | 64 | 1.6410256 | 0.973009447 |
| Fabric Mask | 131 | | 200 | 1.5267176 | 1.097357604 |

| ANOVA | | | | Not Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 4.442173412 | 4 | 1.1105434 | 1.149720874 | 0.332538315 | 2.392164 |
| Within Groups | 425.9726248 | 441 | 0.9659243 | | | |
| Total | 430.4147982 | 445 | | | | |

# Q10. The mask did not leave traces or marks on my face during continuous use.

**DATA: Summary** 

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 100 | 156 | 21 | 39 | 133 |
| Average | 2.2 | 1.6 | 2.7 | 2.3 | 1.6 |
| Mode | 1 | 1 | 1 | 2 | 1 |
| Median | 2 | 1 | 2 | 2 | 1 |
| SD | 1.36 | 0.87 | 1.49 | 1.15 | 1.00 |

## **ANOVA: Single Factor**

**SUMMARY** 

| Groups | Count | Sum | Average | Variance |
|---------------|-------|-----|-----------|-------------|
| Focal Mask | 100 | 222 | 2.22 | 1.85010101 |
| Surgical Mask | 156 | 243 | 1.5576923 | 0.751488834 |
| N95 | 21 | 56 | 2.6666667 | 2.233333333 |
| KN95 | 39 | 91 | 2.3333333 | 1.333333333 |
| Fabric Mask | 133 | 216 | 1.6240602 | 1.009113693 |

| ANOVA | | | | Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 56.90974961 | 4 | 14.227437 | 11.95996965 | 3.07701E-09 | 2.392027 |
| Within Groups | 528.1771101 | 444 | 1.1895881 | | | |
| Total | 585.0868597 | 448 | | | | |

Bonferroni correction:

0.005

## **Bonferroni Post Hoc Test (t-test)**

| | P Value | Hypothesis |
|------------------------------|-------------|------------|
| Focal Mask vs Surgical Mask | 3.25151E-06 | Alternate |
| Focal Mask vs N95 | 0.181233394 | Null |
| Focal Mask vs KN95 | 0.646595644 | Null |
| Focal Mask vs Fabric Mask | 0.00015451 | Alternate |
| Surgical Mask vs N95 | 1.57304E-06 | Alternate |
| Surgical Mask vs KN95 | 6.00014E-06 | Alternate |
| Surgical Mask vs Fabric Mask | 0.54705372 | Null |
| N95 vs KN95 | 0.340747469 | Null |
| N95 vs Fabric Mask | 6.58872E-05 | Alternate |
| KN95 vs Fabric Mask | 0.000246495 | Alternate |

# Q11. The mask stayed away from my lips when I had it on.

#### **DATA: Summary**

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 100 | 156 | 21 | 39 | 133 |
| Average | 1.5 | 2.4 | 1.9 | 1.7 | 2.6 |
| Mode | 1 | 3 | 1 | 1 | 3 |
| Median | 1 | 2.5 | 1 | 1 | 3 |
| SD | 0.72 | 0.99 | 1.28 | 1.02 | 1.07 |

## **ANOVA: Single Factor**

**SUMMARY** 

| Groups | Count | Sum Average | | Variance |
|---------------|-------|-------------|-----------|-------------|
| Focal Mask | 100 | 148 | 1.48 | 0.514747475 |
| Surgical Mask | 156 | 382 | 2.4487179 | 0.984449959 |
| N95 | 21 | 39 | 1.8571429 | 1.628571429 |
| KN95 | 39 | 67 | 1.7179487 | 1.049932524 |
| Fabric Mask | 133 | 344 | 2.5864662 | 1.153451811 |

| ANOVA | | | | Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 92.75025173 | 4 | 23.187563 | 24.03898439 | 5.09835E-18 | 2.392027 |
| Within Groups | 428.2742472 | 444 | 0.9645816 | | | |
| Total | 521.0244989 | 448 | | | | |

Bonferroni correction:

0.005

## **Bonferroni Post Hoc Test (t-test)**

| | P Value | Hypothesis |
|------------------------------|-------------|------------|
| Focal Mask vs Surgical Mask | 2.32643E-15 | Alternate |
| Focal Mask vs N95 | 0.063202005 | Null |
| Focal Mask vs KN95 | 0.124000173 | Null |
| Focal Mask vs Fabric Mask | 1.52934E-16 | Alternate |
| Surgical Mask vs N95 | 0.014305624 | Null |
| Surgical Mask vs KN95 | 6.3984E-05 | Alternate |
| Surgical Mask vs Fabric Mask | 0.647184867 | Null |
| N95 vs KN95 | 0.647184867 | Null |
| N95 vs Fabric Mask | 0.005497158 | Null |
| KN95 vs Fabric Mask | 1.3312E-05 | Alternate |

# Q12. The mask did not have an odor to it when I wore it.

**DATA: Summary** 

| | Focal Mask | Surgical Mask | N95 | KN95 | Fabric Mask |
|---------|------------|---------------|------|------|-------------|
| Count | 100 | 156 | 21 | 39 | 133 |
| Average | 1.7 | 1.9 | 2.1 | 2.3 | 2.2 |
| Mode | 1 | 1 | 2 | 2 | 1 |
| Median | 1 | 2 | 2 | 2 | 2 |
| SD | 0.98 | 0.94 | 1.15 | 1.23 | 1.08 |

## **ANOVA: Single Factor**

**SUMMARY** 

| Groups | Count | Sum Average | | Variance |
|---------------|-------|-------------|-----------|-------------|
| Focal Mask | 100 | 173 | 1.73 | 0.966767677 |
| Surgical Mask | 156 | 292 | 1.8717949 | 0.886683209 |
| N95 | 21 | 45 | 2.1428571 | 1.328571429 |
| KN95 | 39 | 88 | 2.2564103 | 1.511470985 |
| Fabric Mask | 133 | 295 | 2.2180451 | 1.156641604 |

| ANOVA | | | | Significant | | |
|---|---|---|---|---|---|---|
| Source of Variation | SS | df | MS | F | P-value | F crit |
| Between Groups | 19.11440554 | 4 | 4.7786014 | 4.515887444 | 0.001383746 | 2.392027 |
| Within Groups | 469.8299152 | 444 | 1.0581755 | | | |
| Total | 488.9443207 | 448 | | | | |

Bonferroni correction:

0.005

## **Bonferroni Post Hoc Test (t-test)**

| | P Value | Hypothesis |
|------------------------------|-------------|------------|
| Focal Mask vs Surgical Mask | 0.249041242 | Null |
| Focal Mask vs N95 | 0.092363983 | Null |
| Focal Mask vs KN95 | 0.009323133 | Null |
| Focal Mask vs Fabric Mask | 0.000456858 | Alternate |
| Surgical Mask vs N95 | 0.229985486 | Null |
| Surgical Mask vs KN95 | 0.033774254 | Null |
| Surgical Mask vs Fabric Mask | 0.003801344 | Alternate |
| N95 vs KN95 | 0.728655841 | Null |
| N95 vs Fabric Mask | 0.768502087 | Null |
| KN95 vs Fabric Mask | 0.849920213 | Null |